CLINICAL TRIAL: NCT00304525
Title: A Phase I/II, Open-label, Dose Escalation Trial to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of RAF265 (CHIR-265)Administered Orally to Patients With Locally Advanced or Metastatic Melanoma.
Brief Title: A Study to Evaluate RAF265, an Oral Drug Administered to Subjects With Locally Advanced or Metastatic Melanoma
Acronym: CHIR-265-MEL01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRAF265A2101; 2007-005367-10 (EudraCT Number); NCT00324935 (obsolete NCT alias)
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-08

CONDITIONS: Metastatic Melanoma
Keywords: Anti-angiogenesis therapy; Kinase inhibitor therapy; Raf inhibitor; Locally Advanced Melanoma
MeSH Terms: conditions — Melanoma | interventions — RAF265

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- RAF265 - Arm 1 (Experimental): Patients received 10mg RAF265 as a once weekly dose until progressive disease was confirmed.
  Interventions: Drug: RAF265
- RAF265 - Arm 2 (Experimental): RAF265 is given as a single "PK run-in" dose, a single loading dose on day 1 of cycle 1, followed by once daily maintenance doses.
  Interventions: Drug: RAF265
- RAF265 - Arm 3 (Experimental): Patients were treated with once weekly dosing of RAF265
  Interventions: Drug: RAF265
- RAF265 - Arm 4 (Experimental): Patients with locally advanced or metastatic melanoma will utilize a dose close to or at the MTD/RPTD of the liquid formulation that was determined in Arm 2.
  Interventions: Drug: RAF265
- RAF265 - Arm 5 (Experimental): RAF265 was administered as a continuous dose for 2 weeks followed by a dose holiday of 1 week.
  Interventions: Drug: RAF265

INTERVENTIONS:
Drug: RAF265 — A liquid nonaqueous oral formulation. Switched to a tablet formulations with was 60% bioavailable, relative to the liquid at 50mg dose. The liquid dose will be multiplied by a factor of 1.67 to achieve a comparable tablet dose. Tablets are available in 10mg and 50mg strengths.

SUMMARY:
The purpose of this study is to determine the safety profile, pharmacokinetics, pharmacodynamics and maximum tolerated dose of RAF265 in patients with locally advanced and metastatic melanoma.

Phase II portion of study (dose expansion) has been cancelled with Amendment 7 as of Dec 2011.

DETAILED DESCRIPTION:
The Ras/Raf/MEK/ERK pathway plays a prominent role in controlling several key cellular functions including growth, proliferation and survival. B-Raf is a member of the Ras/Raf/MEK/ERK pathway and is frequently mutated in melanoma resulting in activation of the MAPK pathway. RAF265 is a novel, orally active, small molecule with potent inhibitory activity against B-Raf kinase and additional antiangiogenic activity through inhibition of vascular endothelial growth factor receptor type 2 (VEGFR-2) in non-clinical studies.

The primary objectives of this study are to determine the maximum tolerated dose (MTD), dose limiting toxicities (DLTs), and the safety profile of RAF265 when administered orally to subjects with locally advanced or metastatic melanoma; to determine the plasma pharmacokinetics (PKs) of orally administered RAF265; and to evaluate potential pharmacodynamic effects of RAF265 using tumor biopsies, peripheral blood samples, and tumor imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of melanoma, locally advanced AJCC Stage IIIB to metastatic Stage IV
2. Measurable disease - at least one lesion measured in at least one dimension as ≥ 20 mm with conventional techniques or ≥ 10 mm with spiral computed tomography (CT) scan
3. ECOG performance status of 0 or 1
4. No concurrent anticancer or investigational therapy for at least 4 weeks prior to enrollment
5. No major surgery for at least 4 weeks prior to enrollment

Exclusion Criteria:

1. Significant cardiac disease or other significant medical/psychiatric disease
2. History of primary central nervous system tumor or brain metastases
3. History of melena, hematemesis, or hemoptysis within the last 3 months
4. Previous therapy with certain molecularly targeted agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2006-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | at the end of dose escalation
Dose limiting toxicities | during the PK run-in phase and first cycle (28 day cycle)
Safety profile | throughout the study
Evaluate potential pharmacodynamic effects | throughout the study
Pharmacokinetic profile | throughout the study

SECONDARY OUTCOMES:
Evaluate whether somatic mutations in BRAF and N-RAS genes are associated with modulation of pharmacodynamic markers and clinical response | throughout the study
Determine the response rate for BRAF mutant patients | Every 2 months
Determine the recommended phase two dose | at the end of dose escalation

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (11):
- United States (10):
  - University of Colorado Univ.ofColoradoCancerCenter, Aurora, Colorado
  - Georgia Regents University Cancer Clinical Research Unit, Augusta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center/Johns Hopkins Med. Medical Oncology, Baltimore, Maryland
  - Massachusetts General Hospital Dept of Cancer for Melanoma, Boston, Massachusetts
  - Dana Farber Cancer Institute DFCI, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center Dept.ofBethIsraelDeaconess(3), Boston, Massachusetts
  - University of Pennsylvania Health System Dept of Hospital of UnivofPenn, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute Dept of Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center Dept. of Cancer Center, Nashville, Tennessee
  - University of Texas/MD Anderson Cancer Center Onc. Dept,, Houston, Texas
- Novartis Investigative Site, Zurich, Switzerland

REFERENCES:
- See also: CRAF265A2101 Results at Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13806